CLINICAL TRIAL: NCT04852315
Title: Effects of Acute Caffeine Ingestion on Futsal Performance in Sub-elite Players
Brief Title: Acute Caffeine Ingestion on Futsal Performance
Acronym: CAFFFUTSAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Universidad Miguel Hernandez de Elche (Other); University of Beira Interior (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidad Francisco Vitoria
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Caffeine; Placebo
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine supplementation (Experimental): Acute caffeine supplementation
  Interventions: Dietary Supplement: Caffeine
- Placebo supplementation (Placebo Comparator): Acute placebo supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Gelatine capsule with caffeine (3 mg/kg body mass of caffeine) (Bulk Powders, London, United Kingdom). The capsule containing the treatment was ingested with 150 mL of water 60 minutes before the onset of the experiment to allow substance absorption.
  Arms: Caffeine supplementation
Dietary Supplement: Placebo — Gelatine capsule with placebo (Cellulose; Guinama, Valencia, Spain). The capsule containing the treatment was ingested with 150 mL of water 60 minutes before the onset of the experiment to allow substance absorption.
  Arms: Placebo supplementation

SUMMARY:
Caffeine supplementation has been recognized such as an useful strategy for improving performance in intermittent sports, however caffeine ingestion in futsal has been barely studied. In this randomized placebo-controlled study, we investigated the effects of acute caffeine supplementation in improving neuromuscular performance and physical match activity in futsal players.

DETAILED DESCRIPTION:
To date, no previous investigation has studied the effect of acute caffeine ingestion on futsal performance during futsal-specific testing and during a simulated match. Therefore, the aim of this investigation was to establish the effects of acute caffeine intake on futsal-specific tests (e.g. futsal kicking velocity) and match-play running performance in male futsal players.

ELIGIBILITY:
Inclusion Criteria:

* Sub-elite men futsal players

Exclusion Criteria:

* Intolerance to caffeine,
* Suffering from any chronic pathology or an injury in the month prior to the investigation
* Use of medicines or dietary supplements during the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Changes in futsal match-play demands (m/min) | 48-hours
  Using a wireless inertial movement unit system

SECONDARY OUTCOMES:
Changes in maximal jump height (cm) | 48-hours
  Infrared beam jump system
Changes in 20-m sprint test (s) | 48-hours
  Time to complete 10-m and 20-m sprints using photocell timing gates
Futsal kicking velocity and accuracy test (km/h) | 48-hours
  Throwing velocity using a radar gun

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro L López Samanes, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Samanes A, Moreno-Perez V, Travassos B, Del Coso J. Effects of acute caffeine ingestion on futsal performance in sub-elite players. Eur J Nutr. 2021 Dec;60(8):4531-4540. doi: 10.1007/s00394-021-02617-w. Epub 2021 Jun 16. PMID 34132880